CLINICAL TRIAL: NCT02139189
Title: RESTORE Myocardial Function With CorMatrix® ECM® Particulate (P-ECM) Implantation in Subjects With LVEF 25 to 40% Study
Brief Title: Restore Myocardial Function With CorMatrix® ECM® Particulate (P-ECM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corvivo Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-PR-1083
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P-ECM Implant (Experimental): P-ECM Implant into damaged ischemic and/or infarcted myocardium
  Interventions: Device: P-ECM Implant

INTERVENTIONS:
Device: P-ECM Implant — P-ECM Implant into damaged ischemic and/or infarcted myocardium

SUMMARY:
The purpose of this CorMatrix P-ECM safety and feasibility study is to evaluate the safety and functional effect of the CorMatrix P-ECM.

DETAILED DESCRIPTION:
Evaluate the safety of the CorMatrix ECM Particulate (P-ECM) delivered trans-epicardially to subjects with left ventricular ejection fraction (LVEF) 25 to 40% during coronary artery bypass grafting (CABG)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years of age
* Ischemic cardiomyopathy with LVEF 25 to 40% as determined by resting cardiac echocardiography
* Subjects with severe chronic ischemic cardiomyopathy manifested by Canadian Cardiovascular Society (CCS) class II or greater angina, and/or New York Heart Association (NYHA) class II or greater dyspnea
* Patients who have undergone diagnostic coronary angiography demonstrating > 70% diameter narrowing of at least two major coronary arteries or branches OR > 50% diameter narrowing of the left main coronary artery
* Significant left ventricular systolic dysfunction evaluated by echocardiography or LV angiography (LVEF 25 to 40%) due to a prior myocardial infarction. This area of left ventricular dysfunction should be akinetic or severely hypokinetic, not aneurysmal, when assessed by echocardiography or LV angiogram

Exclusion Criteria:

* Need for urgent or emergent revascularization
* Patients with confirmed myocardial infarction within 14 days, and/or rising cardiac biomarker proteins (i.e., CK-MB or troponin), and/or worsening ECG changes
* Patient supported by balloon pump pre-op
* Moderate or severe (> 1+) aortic insufficiency as determined by echocardiogram
* History of severe ventricular tachyarrhythmias requiring treatment
* Hypertrophic obstructive cardiomyopathy (HOCM), restrictive cardiomyopathy, or congenital heart disease
* Prior cardiac operations
* Anticipated for concomitant surgical procedure at the time of CABG (e.g., valve repair or replacement, aneurysm resection, carotid endarterectomy, etc.)
* Active infection, with a temperature greater than 37.5°C and an unexplained white blood cell count in excess of 15,000/mm3 within 48 hours prior to surgery
* Hemoglobin less than 10g/dL, white blood cell count less than 4,000/mm3, absolute neutrophil count less than 1500/mm3
* Primary coagulopathy or platelet disorder, including thrombocytopenia with absolute platelet count < 80k or active state of disseminated intravascular coagulation
* Hemodynamically unstable patients, as defined by heart rate <40/min or >100/min, and/or systolic blood pressure <90 mmHg or >200 mmHg, and/or ongoing need for intravenous inotropic or vasopressor medications
* Severe pulmonary hypertension as defined by PVR > 8 Wood units, that is unresponsive to vasodilator therapy within 14 days of enrollment
* History of stroke or a history of cerebral vascular disease with significant (> 80%) extra cranial stenosis, without evidence of collateral flow. (Patients with cerebral vascular disease history must have acceptable stenosis documented by a carotid doppler study)
* Severe chronic renal insufficiency (serum creatinine >2.5mg/dl, estimated glomular filtration rate (eGFR) <35 mL/min/1.73m2 or need for dialysis)
* Evidence of intrinsic hepatic disease as defined as liver enzyme values (AST or ALT or total bilirubin) that are > 5 times the upper limit of normal within 30 days of enrollment (diagnosis of cirrhosis, chronic hepatitis), except in association with acute decompensation as determined by the Investigator
* Significant peripheral vascular disease defined by claudication, rest pain or leg ulceration
* Positive laboratory test results or a history of syphilis, Hepatitis B Virus, Hepatitis C Virus, Human T-Lymphotropic Virus Type 1 and 2, and Human Immunodeficiency Virus
* Active or known non-dermatological malignancy undergoing treatment including chemotherapy and radiotherapy or any other condition that would place the patient at increased risk for complications during the first 6 months after the procedure in the judgment of the attending cardiologist or cardiac surgeon
* Immunosuppressive medication (e.g. prednisone, cyclophosphamide, etanercept, etc.)
* Previous solid organ transplantation or anticipated need for solid organ transplant other than heart (with the exception of corneal transplant)
* Hematological disorders (e.g., aplastic anemia) or bone marrow disorders
* Myelodysplastic syndrome
* Any condition associated with a life expectancy of less than 6 months
* Contraindications to magnetic resonance imaging (MRI) including presence of an implantable cardiac defibrillator (ICD) or permanent pacemaker (PPM), or cases in which it is anticipated that an ICD or PPM will be implanted prior to the 6 month follow-up or claustrophobia (thus precluding performance of follow-up MRI scans)
* Contraindication to the administration of heparin, warfarin or anti-platelet agents
* Known allergic reaction or sensitivity to porcine material
* Significant cognitive impairment or psychiatric disease (including drug or alcohol abuse) that is likely to impair compliance with the study protocol
* Current participation or participation within the last 3 months in the study of an investigational drug, device, or biologic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Subject-level incidence of serious adverse device effects (SADEs) or serious implantation procedure-related adverse events that occur within 6 months of implantation of the P-ECM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Suwalski, Professor, Principal Investigator — Central Clinical Hospital of the Ministry of Interior in Warsaw
Locations (1):
- Central Clinical Hospital of the Ministry of the Interior in Warsaw, Warsaw, Poland